CLINICAL TRIAL: NCT07162792
Title: The Safety and Efficacy of New-Generation Bioabsorbable Scaffolds Versus Drug-Coated Balloons in the Treatment of De Novo Lesions in Large Coronary Arteries: A Prospective Randomized Controlled Study
Brief Title: The Safety and Efficacy of New-Generation BRS vs. DCB for De Novo Large Coronary Artery Lesions: A Prospective RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-02-011-H01
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease(CAD); de Novo Coronary Lesions
Keywords: drug-coated balloon; percutaneous coronary intervention; bioresorbable scaffold
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRS group (Experimental)
  Interventions: Device: bioresorbable scaffold
- DCB group (Experimental)
  Interventions: Device: drug-coated balloon

INTERVENTIONS:
Device: bioresorbable scaffold — 75 subjects with de novo large vessel coronary lesions who met the inclusion/exclusion criteria were enrolled; subjects were assigned to the treatment group of BRS.
  Arms: BRS group
Device: drug-coated balloon — 75 subjects with de novo large vessel coronary lesions who met the inclusion/exclusion criteria were enrolled; subjects were assigned to the treatment group of DCB.
  Arms: DCB group

SUMMARY:
This study plans to enroll 150 patients who are candidates for "intervention without implantation" therapy and they will be randomly assigned in a 1:1 ratio to either the new-generation Firesorb scaffold group (BRS group, N=75) or the drug-coated balloon group (DCB group, N=75). All enrolled patients will undergo angiographic follow-up at 1 year post-procedure, and serial follow-up (via telephone or outpatient visit) will be performed at 1 month, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years post-procedure. The primary study endpoint was percentage diameter stenosis at 1 year post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* - Radiography inclusion criteria

  1. angiographically confirmed de novo coronary artery lesion;
  2. target lesion stenosis must be ≥70% or ≥50% with clear evidence of myocardial ischaemia (visual assessment);
  3. target lesion vessel diameter is between 2.75mm and 4.0mm, target lesion length must be ≤25mm (visual assessment);
  4. either one or two target lesions to be treated; if two target lesions, they must be located in different target vessels;
  5. successful target lesion preparation: residual stenosis ≤30%, no flow-restricting entrapment, and TIMI grade 3 flow; General inclusion criteria

  <!-- -->

  1. subjects at the age between ≥18 and ≤80 years old;
  2. patients with symptoms or evidence of myocardial ischaemia;
  3. subjects are willing to participate in the study, sign informed consent form, and accept clinical follow-up after operation.

Exclusion Criteria:

* 1. in-stent lesions; 2. For the left main disease, chronic total occlusive lesions; 3. bifurcation lesion (reference vessel diameter of side branch vessels > 2.0 mm); 4. Severely calcified lesions and tortuous lesions; lesions that have failed pretreatment; lesions unsuitable for balloon delivery and dilatation; 5. Previous use of any brand of drug-coated balloon in the target vessel. General inclusion criteria

  1. Any patient with myocardial infarction within one month;
  2. Patients with severe congestive heart failure (NYHA Level III severe heart failure) or severe valvular heart disease; or left ventricular ejection fraction of less than 40%;
  3. Patients with stroke, peptic ulcer or gastrointestinal bleeding within the past 6 months; or patients with bleeding tendency or coagulation disorders;
  4. Patients with severe liver failure (ALT and AST are larger than 3 times of the upper limit of normal value), who are judged to be not applicable to angiography by investigators;
  5. Patients with severe renal failure(eGFR<30ml/minute) or such medical history, failure to comply with angiography conditions;
  6. Subjects who are intolerance or allergic to heparin, contrast agent, polyethylene oxide and polylactic acid - glycolic acid polymer;
  7. Patients who plans to accept selective operation within 1 year;
  8. Patients who are participating in the clinical trial of other drug or device without reaching the time limit of primary endpoint;
  9. Subjects who are considered to be not applicable to be enrolled by investigators due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-23 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
percentage diameter stenosis | 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yerasi C, Case BC, Forrestal BJ, Torguson R, Weintraub WS, Garcia-Garcia HM, Waksman R. Drug-Coated Balloon for De Novo Coronary Artery Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Mar 10;75(9):1061-1073. doi: 10.1016/j.jacc.2019.12.046. PMID 32138967
- [Background] Salloum E, Ohri A, Bartlett F, Ivey T, Savona S. Priapism in sickle cell disease: possible contributory effect of cocaine use. Arch Intern Med. 1993 Oct 11;153(19):2287. No abstract available. PMID 8215732
- [Background] Gauthier BM, Hickner JM, Ornstein S. High prevalence of overweight children and adolescents in the Practice Partner Research Network. Arch Pediatr Adolesc Med. 2000 Jun;154(6):625-8. doi: 10.1001/archpedi.154.6.625. PMID 10850513
- [Background] Yu X, Wang X, Ji F, Zhang W, Yang C, Xu F, Wang F. Correction to: A Non-inferiority, Randomized Clinical Trial Comparing Paclitaxel-Coated Balloon Versus New-Generation Drug-Eluting Stents on Angiographic Outcomes for Coronary De Novo Lesions. Cardiovasc Drugs Ther. 2022 Dec;36(6):1261-1262. doi: 10.1007/s10557-021-07183-1. No abstract available. PMID 33842993
- [Background] Wang Z, Yin Y, Li J, Qi W, Yu B, Xu Z, Zhu W, Yang F, Cao M, Zhang H. New Ultrasound-Controlled Paclitaxel Releasing Balloon vs. Asymmetric Drug-Eluting Stent in Primary ST-Segment Elevation Myocardial Infarction - A Prospective Randomized Trial. Circ J. 2022 Mar 25;86(4):642-650. doi: 10.1253/circj.CJ-21-0315. Epub 2021 Nov 10. PMID 34759131
- [Background] Vos NS, Amoroso G, Herrman JR, Patterson MS, van der Schaaf RJ, Slagboom T, Vink MA. Pronounced late acquired focal coronary artery dilatation after paclitaxel-coated balloon angioplasty: observations from the randomized REVascularization With PaclitaxEL-Coated Balloon Angioplasty Versus Drug-Eluting Stenting in Acute Myocardial InfarcTION (REVELATION) trial. Coron Artery Dis. 2022 Mar 1;33(2):151-152. doi: 10.1097/MCA.0000000000001047. No abstract available. PMID 35112669
- [Background] Shin ES, Lee JM, Her AY, Chung JH, Eun Lee K, Garg S, Nam CW, Doh JH, Koo BK. Prospective randomized trial of paclitaxel-coated balloon versus bare-metal stent in high bleeding risk patients with de novo coronary artery lesions. Coron Artery Dis. 2019 Sep;30(6):425-431. doi: 10.1097/MCA.0000000000000755. PMID 31009399
- [Background] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115
- [Background] Nishiyama N, Komatsu T, Kuroyanagi T, Fujikake A, Komatsu S, Nakamura H, Yamada K, Nakahara S, Kobayashi S, Taguchi I. Clinical value of drug-coated balloon angioplasty for de novo lesions in patients with coronary artery disease. Int J Cardiol. 2016 Nov 1;222:113-118. doi: 10.1016/j.ijcard.2016.07.156. Epub 2016 Jul 27. PMID 27494722
- [Background] Gobic D, Tomulic V, Lulic D, Zidan D, Brusich S, Jakljevic T, Zaputovic L. Drug-Coated Balloon Versus Drug-Eluting Stent in Primary Percutaneous Coronary Intervention: A Feasibility Study. Am J Med Sci. 2017 Dec;354(6):553-560. doi: 10.1016/j.amjms.2017.07.005. Epub 2017 Jul 19. PMID 29208251